CLINICAL TRIAL: NCT06022354
Title: A Single-center, Randomized, Double-blind, Sponsor Open, Placebo-controlled, Dose-escalation Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SIM0278 After Single and Multiple Subcutaneous Injections in Chinese Healthy Subjects
Brief Title: To Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SIM0278 in Chinese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIM0278-101
Record Dates: First submitted 2023-08-15; First posted 2023-09-01 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Part 1 : cohort 1: SIM0278 or placebo (Experimental)
  Interventions: Drug: SIM0278 Injection/Placebo
- Part 1 : cohort 2: SIM0278 or placebo (Experimental)
  Interventions: Drug: SIM0278 Injection/Placebo
- Part 1 : cohort 3: SIM0278 or placebo (Experimental)
  Interventions: Drug: SIM0278 Injection/Placebo
- Part 1 : cohort 4: SIM0278 or placebo (Experimental)
  Interventions: Drug: SIM0278 Injection/Placebo
- Part 1 : cohort 5: SIM0278 or placebo (Experimental)
  Interventions: Drug: SIM0278 Injection/Placebo
- Part 1 : cohort 6: SIM0278 or placebo (Experimental)
  Interventions: Drug: SIM0278 Injection/Placebo
- Part 1 : cohort 7: SIM0278 or placebo (Experimental)
  Interventions: Drug: SIM0278 Injection/Placebo
- Part 2 : cohort 1: SIM0278 or placebo (Experimental)
  Interventions: Drug: SIM0278 Injection/Placebo
- Part 2 : cohort 2: SIM0278 or placebo (Experimental)
  Interventions: Drug: SIM0278 Injection/Placebo
- Part 2 : cohort 3: SIM0278 or placebo (Experimental)
  Interventions: Drug: SIM0278 Injection/Placebo
- Part 2 : cohort 4: SIM0278 or placebo (Experimental)
  Interventions: Drug: SIM0278 Injection/Placebo

INTERVENTIONS:
Drug: SIM0278 Injection/Placebo — SIM0278 Injection/Placebo

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled trial of SIM0278 in healthy subjects. The study will be conducted in 2 parts. Part 1 is single ascending dose study. Part 2 is multiple ascending dose study.

DETAILED DESCRIPTION:
The study will assess the safety, tolerability, and pharmacokinetics（PK） after a single or multiple administration of SIM0278 or placebo via subcutaneous injection in healthy subjects (male or female) where PK, pharmacodynamics (PD) and biomarkers will be assessed. Approximately 68 subjects (up to 84) will be enrolled in the whole study. The ratio of active drug to placebo in each dose level will be 3:1. In part1, approximately 44 subjects (up to 52) will be enrolled for the single dose escalation. Six dose levels are planned in part 1. In part2, approximately 24 (up to 32) subjects will be enrolled for the multiple dose escalation. Three dose levels are planned in part 2.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be 18 to 55 years of age (inclusive), at the time of signing the informed consent.
2. Body Mass Index (BMI) ≥ 18 and ≤ 28 kg/m2 and weight at least 45 kg at screening.
3. A condition of general good health, as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, vital signs, laboratory profile, a 12-lead electrocardiogram (ECG) and chest X-ray.
4. A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   * Not a woman of childbearing potential (WOCBP) as defined in, OR
   * A WOCBP who agrees to follow the contraceptive guidance in from screening through at least 90 days after the last dose of study drug; a WOCBP must have a negative beta-human chorionic gonadotropin (β-hCG) test at screening and baseline prior to administration of investigational product.
5. A male subject must agree to use contraception as detailed in this protocol from screening through at least 90 days after the last dose of study drug. Sperm donation is also restricted during the time-frame that males must practice highly effective method of contraception. This criterion may be waived for male subjects who have had a vasectomy more than (>) 90 days prior to screening.
6. Must voluntarily sign and date each informed consent approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria:

1. History of significant sensitivity to any drug or previous severe adverse reaction to subcutaneous medication.
2. Subject has a history of any clinically significant cardiac, respiratory (including asthma, bronchospasm), renal, hepatic, gastrointestinal, psychiatric, neurologic, hematologic or rheumatic disease, or psychiatric disease or disorder, current acute or chronic infections, or other abnormality that may affect safety, or potentially influence the study results, judged by the investigator.
3. Chronic or active infection(s) requiring treatment with intravenous anti-infectives within 4 weeks prior to the dose of study drug, or oral anti-infectives within 2 weeks prior to Day 1, or positive test for novel coronavirus antigen or nucleic acid within 4 weeks prior to first dose
4. Evidence or history of malignancy other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma.
5. History of chronic or active hepatitis, or current positive result, including hepatitis B or hepatitis C infection, as evidenced by a positive test for hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody (HCV Ab).
6. History of tuberculosis (TB), or active or latent TB on the basis of positive medical history.
7. History of or positive screening test for human immunodeficiency virus (HIV) infection; any genetic, congenital, or acquired immunodeficiency syndrome, or any chronic recurring infections (including mucocutaneous candidiasis).
8. Systolic blood pressure (BP) ≥ 140 mmHg or ≤ 90 mmHg, or diastolic BP≥ 90 mmHg or ≤50 mm Hg, or HR > 100 bpm, at Screening or baseline，and abnormal clinically significant should be judged by the investigator
9. Subjects with ANY of the following abnormalities in clinical laboratory tests at screening:

   * Neutrophil or lymphocyte counts below the normal range; Eosinophil count above the normal range.
   * Estimated glomerular filtration rate (GFR) by Chronic Kidney Disease Epidemiology Collaboration equation (CKD-EPI) calculation ≤90 mL/min/1.73 m2 at screening.
   * Aspartate aminotransferase (AST)、Alanine transaminase (ALT) >1.5 x upper limit of normal (ULN)
   * Total bilirubin >1.2 x ULN
   * Other clinically significant abnormalities of laboratory assessments, as judged by the Investigator and/or sponsor Medical Monitor, that could affect the safety of the subject, or the interpretation of the data from the study.
10. 12-lead ECG demonstrating QTcF≥450 msec（male）or QTcF≥470 msec（female） at Screening. Subject who have II or III degree atrioventricular block or other clinically significant electrocardiogram abnormalitieshas, in the opinion of the investigator, are unsuitable subjects in the study.
11. Use of prescription or non-prescription drugs (including recreational drugs and herbal medications) within 14 days or 5 half-lives (whichever is longer) prior to Day 1 and/or within the duration of the study.
12. Treatment with biologic agents (such as monoclonal antibodies including marketed drugs) within 12 weeks or 5 half-lives (whichever is longer) prior to Day 1.
13. Prior administration of any IL-2 based product.
14. Exposure to immune-modulating medications (including topical or systemic use of corticosteroids) within 4 weeks prior to Day 1.
15. Receipt of any investigational product within 3 months or 5 half-lives (whichever is longer) prior to Day 1.
16. Will have live vaccine or attenuated live vaccine shots within the 12 weeks prior to Day 1, or planning to receive these vaccines at any time during study period or within 8 weeks after last dose.
17. Current or history of regular alcohol abuse（14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine）within 6 months prior to day 1. OR Positive screen for alcohol breath test during screening period.
18. Take more than 10 cigarettes/day within the last 3 months prior to day 1, and/or unwilling to stop using any tobacco products during the study duration.
19. History of substance abuse, or a positive urine drug screen within 5 years prior to Screening, or urine drug screening result is positive.
20. Donation or loss of 400 mL or more blood volume (including plasmapheresis) or receipt of a transfusion of any blood product within 8 weeks prior to Day 1.
21. Consideration by the investigator, for any reason, that the subject is an unsuitable candidate to enroll this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) of subcutaneous injections of SIM0278 in healthy subjects after single dose (Part 1) or multiple dose (Part 2) administration | Part 1:up to 29 days after the first dose of treatment; Part 2:up to 85 days after the first dose of treatment

SECONDARY OUTCOMES:
Peak plasma concentration(Cmax) of SIM0278 in serum | Time Frame: Part 1:up to 29 days after the first dose of treatment; Part 2:up to 57 days after the first dose of treatment
  Cmax was measured for SIM0278 administered by subcutaneous injection
Time to reach maximum concentration (Tmax) of SIM0278 in serum | Part 1:up to 29 days after the first dose of treatment; Part 2:up to 57 days after the first dose of treatment
  Tmax was measured for SIM0278 administered by subcutaneous injection
Area under the curve (AUC) of SIM0278in serum | Part 1:up to 29 days after the first dose of treatment; Part 2:up to 57 days after the first dose of treatment
  AUC was measured for SIM0278 administered by subcutaneous injection
Half life (T1/2) of SIM0278 in serum | Part 1:up to 29 days after the first dose of treatment; Part 2:up to 57 days after the first dose of treatment
  T1/2 was measured for SIM0278 administered by subcutaneous injection
Total body clearance (CL/F) of SIM0278 in serum | Part 1:up to 29 days after the first dose of treatment; Part 2:up to 57 days after the first dose of treatment
  CL/F was measured for SIM0278 administered by subcutaneous injection
Total volume of distribution（Vd） at the terminal phase of SIM0278 in serum | Part 1:up to 29 days after the first dose of treatment; Part 2:up to 57 days after the first dose of treatment
  Vd was measured for SIM0278 administered by subcutaneous injection
Incidence of antidrug antibodies (ADA) | Part 1:up to 29 days after the first dose of treatment; Part 2:up to 85 days after the first dose of treatment
  The presence of ADAs to SIM0278 will be listed and summarized by treatment group

OTHER OUTCOMES:
Fold Change from Baseline in Regulatory T cells (Tregs) | Part 1: Pre-dose on Day1 up to 29 days after the first dose of treatment; Part 2: Pre-dose on Day1 up to 71 days after the first dose of treatment
Fold Change from Baseline in Conventional CD4+ T Cells | Part 1: Pre-dose on Day1 up to 29 days after the first dose of treatment; Part 2: Pre-dose on Day1 up to 71 days after the first dose of treatment
Fold Change from Baseline in Conventional CD8+ T Cells | Part 1: Pre-dose on Day1 up to 29 days after the first dose of treatment; Part 2: Pre-dose on Day1 up to 71 days after the first dose of treatment
Fold Change from Baseline in Natural Killer (NK) Cells | Part 1: Pre-dose on Day1 up to 29 days after the first dose of treatment; Part 2: Pre-dose on Day1 up to 71 days after the first dose of treatment
Change from Baseline in Treg Activation Markers: Cytokine Levels, Proliferation and Immunosuppressive Markers Expression | Part 1: Pre-dose on Day1 up to 29 days after the first dose of treatment; Part 2: Pre-dose on Day1 up to 71 days after the first dose of treatment
The correlation between SIM0278 dose/exposure and biomarkers or safety endpoints (if applicable) in healthy subjects | Part 1:up to 29 days after the first dose of treatment; Part 2:up to 71 days after the first dose of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Qingdao University, Qingdao, China, Shandong, China

IPD SHARING:
Plan to Share IPD: No